CLINICAL TRIAL: NCT02794558
Title: A Clinical Study To Evaluate the Safety and Effectiveness of MR Guided Focused Ultrasound Surgery in the Treatment of Early Breast Carcinomas
Brief Title: Safety and Effectiveness of MR Guided Focused Ultrasound Surgery in the Treatment of Early Breast Carcinomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC004
Record Dates: First submitted 2016-06-01; First posted 2016-06-09 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, MRgFus, Focused Ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects in this arm are treated once with MRgFUS device
  Interventions: Device: ExAblate MRgFUS

INTERVENTIONS:
Device: ExAblate MRgFUS — MR images of the breast will be obtained for lesion localization purposes. The breast surgeon or the radiologist will make a treatment plan or map. Sonication at therapeutic power level will be performed on multiple overlapping points successively until sonication of the target volume has been completed.
  Follow-up evaluation will be made within 14 to 21 days after the MRgFUS treatment.
  Other Names: Focused Ultrasound

SUMMARY:
Non-randomized, Single Arm Clinical study to Evaluate the Safety and Effectiveness of MR Guided Focused Ultrasound Surgery in the Treatment of Early Breast Carcinomas

DETAILED DESCRIPTION:
Study specific aim is to Coagulate the tissue volume of a proven breast cancer with MRgFUS and Collect post treatment follow-up clinical and radiological data for a period of 5 years following MRgFUS for breast cancer.

Safety of the treatment will be evaluated by recording and assessing the incidence and severity of device- related complications from the first visit through the 5 years follow-up period.

Secondary objective of this study is to evaluate post treatment local recurrence in the same quadrant or less then 4cm from the periphery of the treated lesion, during a 5 year period following the MRgFUS treatment.

Women with breast cancer in whom breast MR imaging identifies a single focal breast lesion up to 1.5 cm in diameter will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18 years with - breast cancer proven by 14-20 G. core needle biopsy of the breast lesion.
* No evidence of cancer at the sentinel/ Axillary node
* Women in whom breast MR imaging identifies a single focal well-demarcated breast lesion less than or equal to 1.5 cm in diameter with stage T1, N0, M0 disease.
* Patient received neoadjuvant care for 4 weeks such as: Hormone replacement therapy or Tamoxifen is permissible where the tumor is less than or equal to 1.5 before neoadjuvant therapy
* Able and willing to give consent and able to attend all study visits.
* Able to communicate sensations during the MRgFUS procedure.
* Life expectancy of 5 years or more.

Exclusion Criteria:

* Breast cancer which was diagnosed by incisional / excisional biopsy
* Contraindication to MRI (non-MRI compatible implanted metal devices).
* Pregnant or lactating post partum women.
* Prior XRT or laser or cryo-therapy to the target breast.
* Difficulty lying prone and still for up to 210 minutes in the MR unit, e.g., COPD, heart disease, lung disease, sleep apnea or airway problems, severe asthma, severe arthritis, severe claustrophobia.
* Patients with unstable cardiac status including:

  * Unstable angina pectoris on medication.
  * Patients with documented myocardial infarction within six months of protocol entry.
  * Congestive heart failure requiring medication.
  * Patients on anti-arrhythmic drugs.
  * Severe hypertension (diastolic BP > 100 on medication).
  * Patients with cardiac pacemakers.
* Immunosuppressed patients, e.g., patients receiving steroids or other immunosuppressive medication, insulin-dependent diabetes mellitus, collagen vascular disease.
* Patients receiving chemotherapy
* Patients with history of grand mal seizures, severe cerebrovascular disease (multiple CVA or CVA within 6 months), hemolytic anemia (hematocrit < 30), or patients on dialysis.
* Patients currently receiving anticoagulation therapy.
* Large patients who cannot fit comfortably in the magnet, or patients > 100Kg.
* Lesions difficult to target (<1 cm from skin, nipple-areola complex or the ribcage), as visualized on pre-therapy MRI.
* Microcalcifications as the only sign of breast cancer on imaging studies.
* Patients with breast implants.
* Prior reaction to gadolinium-based contrast agent
* Prior radiation to the breast, which is about to be treated.
* Evidence of tumor at any location other then the targeted lesion.
* Histological type of invasive micropapillary carcinoma because of cancer displacement by the needle
* Mucinous carcinoma which was diagnosed by core needle biopsy because of needle cancer displacement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-06; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse events | 5 years
  Safety of the treatment will be evaluated by recording and assessing the incidence and severity of device- related complications

SECONDARY OUTCOMES:
Post treatment local recurrence | 5 years
  new appearance of a malignant tissue of the same type as the treated primary breast lesion, in the same quadrant or less then 4cm from the periphery of the treated lesion, during a 5 year period following the MRgFUS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hidemi Furasawa, MD, Principal Investigator — Managing Director at Breastopia Namba Hospital

IPD SHARING:
Plan to Share IPD: No